CLINICAL TRIAL: NCT05418933
Title: Effects of Family Workshops on Children With Global Developmental Delays and Their Parents
Brief Title: Workshops for Children With Global Developmental Delays
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, MD, Professor, Taipei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKH-111-1
Record Dates: First submitted 2022-06-08; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Global Developmental Delay
Keywords: family workshops
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Family workshops with 5 courses, with 6-7 families in one course, 2 hours per session, one time per week, for a total of 6 weeks.
  Interventions: Other: Family workshop

INTERVENTIONS:
Other: Family workshop — Family workshops for 5 courses, with 6-7 families in one course. The workshops were 2 hours per session, one time per week, for a total of 6 weeks.

SUMMARY:
To investigate the therapeutic effects of family workshops on children with global developmental delays and their parents by the analysis of the previously conducted workshops.

DETAILED DESCRIPTION:
To evaluate the effects of family workshops for children aged 18-36 months old with language developmental delays conducted from Jan 2014 Jan to Dec 2018, by the data analysis.

The participants were children with global developmental delay (language delay with at least one delay in motor, cognitive function, or emotional and social functioning) and their parents in the workshops.

The family workshops were conducted with 5 courses, with 6-7 families in one course, a 2-hour session per week, for 6 weeks.

Effects:

1. Investigate the therapeutic effects of workshops for children with global developmental delays
2. Investigate the therapeutic effects of workshops for the parents of children with global developmental delays

ELIGIBILITY:
Inclusion Criteria:

* Children aged 18-36 months old with global developmental delays (language developmental delay, with motor, cognition, or social and emotional developmental delays) Parents and children attended the one 2 hour-session of workshop per week for 6 weeks

Exclusion Criteria:

* Less than 18 months old or older than 36 months old

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric Outcome Data Collection Instrument | scores change of Pediatric Outcome Data Collection Instrument from baseline to 6 weeks after treatment
  measure the functional performance of children, the minimum and maximum values range from 1 to 100, higher scores mean a better outcome

SECONDARY OUTCOMES:
Mandarin-Chinese Communicative Developmental Inventory | percent change of Mandarin-Chinese Communicative Developmental Inventory from baseline to 6 weeks after treatment
  assess communication function of children, <10% indicates delayed development, 10% or more than 10% indicates normal development
Peabody Developmental Motor Scale | scores change of Peabody Developmental Motor Scale from baseline to 6 weeks after treatment
  assess fine motor function of children, the minimum and maximum values range from 1 to 100, higher scores mean a better outcome
Emotional Competency Rating Scale | scores change of Emotional Competency Rating Scale from baseline to 6 weeks after treatment
  assess the emotional function of children, the minimum and maximum values range from 1 to 100, higher scores mean a better outcome
Pediatric Evaluation of Disability Inventory | scores change of Pediatric Evaluation of Disability Inventory from baseline to 6 weeks after treatment
  assess the functional skill attainment of children, the minimum and maximum values range from 1 to 100, higher scores mean a better outcome
Pediatric Daily Occupation Scale | scores change Pediatric Daily Occupation Scale from baseline to 6 weeks after treatment
  assess the occupational performance in the daily life of children, the minimum and maximum values range from 1 to 100, higher scores mean a better outcome
Pediatric Quality of Life Inventory-Geriatric Core Scale | scores change ofPediatric Quality of Life Inventory-Geriatric Core Scale from baseline to 6 weeks after treatment
  assess the quality of life of children, the minimum and maximum values range from 1 to 100, higher scores mean a better outcome
Pediatric Quality of Life Inventory-Family Impact Module | scores change of Pediatric Quality of Life Inventory-Family Impact Module from baseline to 6 weeks after treatment
  assess the impact of pediatric conditions on family functioning and parental quality of life, the minimum and maximum values range from 1 to 100, higher scores mean a better outcome
Parental satisfaction questionnaire | scores of Parental satisfaction questionnaire after treatment
  assess the parents' satisfaction with the workshops, with scores ranging from 1-to 100, higher scores mean a higher satisfaction
Caregiver Strain Index | scores change of Caregiver Strain Index from baseline to 6 weeks after treatment
  assess family strain, the minimum and maximum values range from 1 to 100, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh WH, Huang PC, Tsai PC, Lee W, Hu Y, Lee WC, Hsieh RL. Short-term multidisciplinary family-centered workshop for preschool children with global developmental delays. Pediatr Res. 2023 Aug;94(2):707-714. doi: 10.1038/s41390-023-02507-3. Epub 2023 Feb 15. PMID 36792650